CLINICAL TRIAL: NCT02352675
Title: Determination of the Minimal Concentration of Antifibrinolytics Required to Inhibit t-PA-activated Fibrinolysis Using an in Vitro Experimental Model of Fibrinolysis.
Brief Title: Determination of the Minimal Concentration of Antifibrinolytics Required to Inhibit t-PA-activated Fibrinolysis
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, David Faraoni, Cardiac Anesthesiologist, Boston Children's Hospital
Other Study IDs: P00016186
Record Dates: First submitted 2015-01-26; First posted 2015-02-02 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Congenital Heart Disease; Fibrinolysis; Rotational Thromboelastometry
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The doctor will obtain one 13.6 mL blood sample from the arterial catheter or intravenous catheter at the beginning of the procedure after the patient has been anesthetized.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Congenital Heart Disease: Infants with congenital heart disease (CHD) who are scheduled to undergo an elective cardiac catheterization lab procedure at Boston Children's Hospital
  Interventions: Other: Intraoperative Blood Sample
- Non Congenital Heart Disease: Infants who do not have congenital heart disease (No-CHD) and are scheduled to undergo a non-cardiac surgery (such as craniofacial surgery, neurosurgery, or orthopedic surgery) in the operating room at Boston Children's Hospital.
  Interventions: Other: Intraoperative Blood Sample

INTERVENTIONS:
Other: Intraoperative Blood Sample — Blood sample will be run using rotational thromboelastometry to determine the minimal concentration of TXA and EACA need to inhibit fibrinolysis

SUMMARY:
Lysine analogs, like tranexamic acid (TXA) or epsilon aminocaproic acid (EACA), are antifibrinolytic agents routinely administered in children undergoing different surgeries associated with a high bleeding risk (e.g. cardiac, craniofacial, and orthopedic surgeries). Although there is a growing literature regarding the pharmacokinetic characteristics of these drugs in children, the plasmatic concentration required to completely inhibit fibrinolysis remains to be determined. In this in vitro study, the investigators will use an experimental model of fibrinolysis designed for rotational thromboelastometry (ROTEM®) to determine the minimal concentration inhibiting fibrinolysis for both TXA and EACA. In addition, this study will be used to create and validate a new experimental assay to measure fibrinolysis and the effect of antifibrinolytic agents.

ELIGIBILITY:
Inclusion Criteria:

* infants between 2 months of age and equal to or less than 12 months of age
* weigh over 5.0 kg
* either have CHD and are scheduled to undergo an elective cardiac catheterization lab procedure or do not have CHD and are scheduled to undergo a non-cardiac surgery (such as craniofacial surgery, neurosurgery, or orthopedic surgery) in the operating room

Exclusion Criteria:

* undergoing an emergent procedure,
* child in a moribund condition (American Society of Anesthesiology (ASA 5)
* children with a hematological and/or oncological disease
* Jehovah witnesses
* children with preoperative coagulopathy, defined as a platelet count < 100,000/μL, fibrinogen level < 100 mg/dL, prothrombin time (PT) and activated partial thromboplastin time (PTT) > 1.5 normal range

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a prospective in vitro study being performed on whole blood obtained from two groups of infants. The first group will include infants with congenital heart disease (CHD) who are scheduled to undergo an elective cardiac catheterization lab procedure at Boston Children's Hospital. The second group will include infants who do not have congenital heart disease (No-CHD) and are scheduled to undergo a non-cardiac surgery (such as craniofacial surgery, neurosurgery, or orthopedic surgery) in the operating room at Boston Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Concentration of antifibrinolytics associated with a complete inhibition of t-PA activated fibrinolysis confirmed by EXTEM test and the Star-TEM test. | One Year

CONTACTS AND LOCATIONS:
Overall Officials: David Faraoni, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Miller BE, Mochizuki T, Levy JH, Bailey JM, Tosone SR, Tam VK, Kanter KR. Predicting and treating coagulopathies after cardiopulmonary bypass in children. Anesth Analg. 1997 Dec;85(6):1196-202. doi: 10.1097/00000539-199712000-00003. PMID 9390579
- [Background] Arnold P. Treatment and monitoring of coagulation abnormalities in children undergoing heart surgery. Paediatr Anaesth. 2011 May;21(5):494-503. doi: 10.1111/j.1460-9592.2010.03461.x. Epub 2010 Dec 1. PMID 21118327
- [Background] Ngaage DL, Bland JM. Lessons from aprotinin: is the routine use and inconsistent dosing of tranexamic acid prudent? Meta-analysis of randomised and large matched observational studies. Eur J Cardiothorac Surg. 2010 Jun;37(6):1375-83. doi: 10.1016/j.ejcts.2009.11.055. Epub 2010 Feb 1. PMID 20117944
- [Background] Eaton MP. Antifibrinolytic therapy in surgery for congenital heart disease. Anesth Analg. 2008 Apr;106(4):1087-100. doi: 10.1213/ane.0b013e3181679555. PMID 18349177
- [Background] Faraoni D, Willems A, Melot C, De Hert S, Van der Linden P. Efficacy of tranexamic acid in paediatric cardiac surgery: a systematic review and meta-analysis. Eur J Cardiothorac Surg. 2012 Nov;42(5):781-6. doi: 10.1093/ejcts/ezs127. Epub 2012 Apr 24. PMID 22531271
- [Background] Faraoni D, Goobie SM. New insights about the use of tranexamic acid in children undergoing cardiac surgery: from pharmacokinetics to pharmacodynamics. Anesth Analg. 2013 Oct;117(4):760-762. doi: 10.1213/ANE.0b013e3182a22278. No abstract available. PMID 24057950
- [Background] Faraoni D. Safety of tranexamic acid in pediatric cardiac surgery: what we do not know. Eur J Cardiothorac Surg. 2011 Dec;40(6):1550-1; author reply 1551-2. doi: 10.1016/j.ejcts.2011.03.009. Epub 2011 Apr 14. No abstract available. PMID 21497106
- [Background] Raza I, Davenport R, Rourke C, Platton S, Manson J, Spoors C, Khan S, De'Ath HD, Allard S, Hart DP, Pasi KJ, Hunt BJ, Stanworth S, MacCallum PK, Brohi K. The incidence and magnitude of fibrinolytic activation in trauma patients. J Thromb Haemost. 2013 Feb;11(2):307-14. doi: 10.1111/jth.12078. PMID 23176206
- [Background] Dekker SE, Viersen VA, Duvekot A, de Jong M, van den Brom CE, van de Ven PM, Schober P, Boer C. Lysis onset time as diagnostic rotational thromboelastometry parameter for fast detection of hyperfibrinolysis. Anesthesiology. 2014 Jul;121(1):89-97. doi: 10.1097/ALN.0000000000000229. PMID 24646494